CLINICAL TRIAL: NCT02187900
Title: Phase 3 Study of Treatment of IgAN With Multi-glycoside of Tripterygium Wilfordii HOOK. f
Brief Title: Treatment of IgAN With Multi-glycoside of Tripterygium Wilfordii HOOK. f.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Youming Peng, Director of the Nephrology Institute, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNXY201401
Record Dates: First submitted 2014-06-22; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: IgA Nephropathy
Keywords: Tripterygium Wilfordii HOOK. f.; Mycophenolate mofetil
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TWH for the treatment of IgAN (Experimental): Interventions :The dosage of 40 mg of Multi-glycoside of Tripterygium Wilfordii HOOK. f. was divided into 2 equal doses at 12-hour intervals for 6 months.
  Interventions: Drug: Multi-glycoside of Tripterygium Wilfordii HOOK. f. (TWH)
- MMF for IgAN (Active Comparator): MMF for the treatment of IgAN for 6 months
  Interventions: Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Multi-glycoside of Tripterygium Wilfordii HOOK. f. (TWH) — The dosage of 40 mg of Multi-glycoside of Tripterygium Wilfordii HOOK. f. was divided into 2 equal doses at 12-hour intervals for 6 months.
  Other Names: Multi-glycoside of Tripterygium Wilfordii HOOK. f.
  Arms: TWH for the treatment of IgAN
Drug: Mycophenolate mofetil (MMF) — Mycophenolate mofetil 1.5mg/day for the treatment of IgAN for 6 months
  Other Names: Mycophenolate mofetil
  Arms: MMF for IgAN

SUMMARY:
The purpose of this study is to determine whether Multi-glycoside of Tripterygium Wilfordii HOOK. f. is effective and safe in the treatment of IgA nephropathy.

DETAILED DESCRIPTION:
Primary IgA nephropathy (IgAN) is the most common form of idiopathic glomerulonephritis throughout of the world. The disease is characterized by the predominant deposition of polymer Gal-deﬁcient IgA1 immune complex（pGd-IgA1-IC）in the glomeruli which leads to the proliferation of mesangial cells. Mycophenolate mofetil is reported to be useful in the treatment of IgAN in Chinese patients, but the price is expensive together with some adverse events. Tripterygium Wilfordii HOOK. f. is a traditional chinese medicine and is useful in the treatment of CKD, the purpose of this study is to determine whether Multi-glycoside of Tripterygium Wilfordii HOOK. f. is effective and safe in the treatment of IgA nephropathy

ELIGIBILITY:
Inclusion Criteria:

* urinary protein levels ≥1.0 g/24 h
* estimated glomerular filtration rate (eGFR) ≥30 ml·min-1·1.73 m-2body surface area by the MDRD formula (eGFR=194×age-0.287×serum creatinine
* 1.094(×0.739, if female) (where sCr is the serum creatinine, dry chemistry method, mg/dl))
* peripheral blood white blood cell count ≥3000×109/L
* no other cause for tubulointerstitial lesions
* no history of immunomodulatory agent intake before renal biopsy
* no systemic infection
* age between 16 and 65 years

Exclusion Criteria:

* severe infections

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-08 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients reaching remission | one year
  (i) complete remission was deﬁned as the absence of proteinuria (24-h urine protein < 0.4 g/24 h), serum albumin >35 g/L and Scr < 1.24 mg/ dL; (ii) partial remission was deﬁned as a 24-h urine protein ≤ 3.5 g/24 h and a decline of >50% of the baseline value with an Scr elevation of <15% of the baseline value; (iii) no response was deﬁned as a 24-h urine protein >3.5 g/24h, or a decline < 50% of base- line value or increase and/or an Scr level >50% of the baseline value

SECONDARY OUTCOMES:
Renal survival | one year
  Renal survival was estimated on the basis of a 50% increase in baseline serum creatinine concentration.

OTHER OUTCOMES:
adverse event | one year
  liver function test result abnormalities;menstrual disturbance

CONTACTS AND LOCATIONS:
Overall Officials: Shenghua Zhou, MD, Study Director — the second xiangya hospital of CSU
Locations (1):
- The second Xiangya Hospital of CSU, Changsha, Hunan, China